CLINICAL TRIAL: NCT03707314
Title: A Randomised Controlled Trial of Very Early Angiography +/- Intervention Versus Standard of Care on Outcomes in Patients With Non ST-elevation Myocardial Infarction
Brief Title: Very Early Versus Delayed Angiography +/- Intervention on Outcomes in Patients With NSTEMI
Acronym: RapidNSTEMI
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Stopped due to low event rate and poor recruitment
Sponsor: University Hospitals, Leicester (Other)
Collaborators: British Heart Foundation (Other); University of East Anglia (Other); University of Leicester (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EDGE 89678
Record Dates: First submitted 2018-07-13; First posted 2018-10-16 (Actual); Last update posted 2022-11-10 (Actual); Status verified 2022-11

CONDITIONS: Cardiovascular; Attack
Keywords: NSTEMI
MeSH Terms: conditions — Non-ST Elevated Myocardial Infarction

STUDY DESIGN:
Intervention Model Description: Multi-centre parallel design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: Immediate angiography (Other): Immediate angiography with follow-on revascularisation if indicated
  Interventions: Procedure: Angiography with follow-on revascularisation if indicated
- Group B: Standard of care angiography (Other): Standard of care angiography with follow-on revascularisation if indicated (within 3-4 days, but will vary depending on recruiting centre)
  Interventions: Procedure: Angiography with follow-on revascularisation if indicated

INTERVENTIONS:
Procedure: Angiography with follow-on revascularisation if indicated — Angiography with follow-on revascularisation (if indicated)

SUMMARY:
Prospective, open, multicentre, randomised controlled trial in patients with higher risk non-ST elevation myocardial infarction acute coronary syndrome

DETAILED DESCRIPTION:
Background: Clinical event rates in Non ST elevation myocardial infarction acute coronary syndrome (N-STEMI ACS) patients remain high, with one year MACE rates as high as 20%. While there may be early mortality differences between N-STEMI and STEMI, outcomes beyond one year become very similar. N-STEMI ACS patients therefore rightly remain the focus of a number of research directives. The objective of the RAPID-NSTEMI trial is to determine if clinical outcomes can be improved by very early intervention in a pre-determined higher risk N-STEMI ACS population. Published data has shown that inpatient Percutaneous Coronary Intervention (PCI) in N-STEMI ACS patients reduces subsequent clinical events. This had led to guidelines supporting its use in clinical practice. However, there is much less certainty regarding the timing of the PCI and, in particular, whether this should be a strategy used early to optimize outcomes. Thus, while evidence based guidelines (NICE and European) provide general time parameters for PCI, immediate angiography with a view to intervention in higher risk patients has never been robustly tested in any adequately powered, prospective randomised trial with clinical end points. The RAPID-NSTEMI trial sets out to test the benefits, or otherwise, of a strategy of immediate angiography with follow-on revascularisation in higher risk N-STEMI ACS patients.

Hypothesis: Very early angiography +/- PCI improves clinical outcomes in higher risk NSTEMI patients when compared to standard invasive management.

Methods: In order to identify higher risk patients as soon as possible after presentation, a high sensitivity troponin (Hs-Troponin-T or Hs-Troponin-I) will be taken, allowing calculation of a GRACE 2.0 score (GS 2.0) early after admission. The GS 2.0 will be determined in sufficient time to be able to test an early intervention strategy arm. Patients with GS 2.0 of ≥118 alone, or ≥90 with additional high risk features will be randomised in a 1:1 fashion to one of two groups:

Group A: immediate angiography with follow-on revascularisation if required Group B: standard care - pharmacological treatment until angiography with follow on revascularisation if required (preferably within 72 hours as per current guidelines).

The primary outcome for the main study will be a 12-month of all-cause mortality, new myocardial infraction and hospital admission with heart failure.

Power calculations indicate that 2314 patients are required to show MACE superiority for early intervention in such higher risk N-STEMI ACS patients.

Analyses will be primarily according to "intention to treat", with a secondary analysis according to trial treatment received (comparing those who actually received follow-on revascularisation at the two different trial time points). There will be a cost effectiveness analysis.

Mechanistic sub-studies in the two groups will be undertaken.

1. Cardiac magnetic resonance imaging substudy to assess differences in infarct size, oedema, microvascular obstruction and left ventricular ejection fraction between the two arms.
2. Novel biomarkers substudy that will be funded separately after appropriate funding applications

Expected value of results: The investigators have designed a superiority trial to anticipate that outcomes will be improved in higher risk patients revascularised very early after presentation with N-STEMI. Irrespective of outcome, this trial should determine whether there is a need for a change in current patient management of a common condition and, in particular, if all N-STEMI patients should be admitted to a PCI-capable hospital to allow for very early intervention. The results will inform national and international guidelines. The planned cost effectiveness analysis will become particularly important if clinical outcomes are no different between groups since length of stay should be different.

ELIGIBILITY:
Inclusion Criteria

* 18 years of age and over
* Patients presenting to hospitals with a clinical diagnosis of non-ST elevation myocardial infarction comprising:

  * Ischaemic symptoms (as defined in Appendix III of protocol)
  * Elevated high sensitivity Troponin T or I (above the normal range for individual hospitals)
* GRACE-2.0 score (www.gracescore.org) of either:

  * ≥118 (corresponding to 6-month death >6%) OR
  * ≥90 but <118 (corresponding to 6-month death >3% but <6%)
* If GRACE 2.0 score ≥90 or <118 must have at least one additional high risk feature:

  * Anterior location of ECG changes (leads V2 - V5)
  * ST-segment depression in 2 contiguous leads (any territory) of 0.15mV/ 1.5mm.
  * Diabetes Mellitus on medication
  * High-sensitivity Troponin I or T 3 x ULN
* Onset of ischaemic symptoms at any time prior to admission but most recent episode within 12 hours to admission
* Intention to perform angiography and, if indicated, follow-on revascularisation
* Provision of assent or written consent
* Randomisation must be performed within 6 hours of admission

Exclusion Criteria

* ST elevation myocardial infarction
* Evident type 2 myocardial infarction (e.g. anaemia)
* Evidence of previous known cardiomyopathy
* Cardiogenic Shock
* Known severe valvular heart disease
* Need for urgent PCI according to ESC Guidelines (haemodynamic instability, VT, VF, recurrent or persistent pain)
* Any contraindication to PCI
* Current participation in another intervention trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 425 (Actual)
Dates: Start 2018-11-06 (Actual); Primary Completion 2021-10-28 (Actual); Study Completion 2021-10-28 (Actual)

PRIMARY OUTCOMES:
Major adverse cardiovascular events | 12 months
  Incidence of the composite of all-cause mortality, new myocardial infarction and admission for heart failure within 12 months following randomisation

SECONDARY OUTCOMES:
All-cause mortality | 12 months
  Incidence of all-cause mortality
New myocardial infarction | 12 months
  Incidence of new myocardial infarction
Heart failure | 12 months
  Incidence of admission for heart failure
Cardiovascular mortality | 12 months
  Incidence of cardiovascular mortality
Length of in-patient stay | Through study completion, 3 years
  Length of in-patient stay (defined as randomisation to first discharge) in days
All-cause mortality prior to planned coronary angiography | During index admission
  Incidence of all-cause mortality prior to planned coronary angiography following index admission with NSTEMI
New myocardial infarction prior to planned coronary angiography | During index admission
  Incidence of new myocardial infarction prior to planned coronary angiography following index admission with NSTEMI
Major bleeding prior to planned coronary angiography | During index admission
  Incidence of major bleeding (classified as BARC 3-5) prior to planned coronary angiography following index admission with NSTEMI
Admission for ischaemia-driven revascularisation | 12 months
  Incidence of admission for ischaemia-driven revascularisation
Admission for any cause | 12 months
  Incidence of admission for any cause
Quality of life measured using Seattle Angina Questionnaire | 12 months
  Quality of life measured using Seattle Angina Questionnaire at 24 hours post procedure, 1 month, 6 months and 12 months
Quality of life measured using EuroQoL-5D-5L questionnaire | 12 months
  Quality of life measured using the EuroQoL-5D-5L questionnaire at 24 hours post procedure, 1 month, 6 months and 12 months
BARC 3-5 bleeding | 12 months
  Incidence of Bleeding Academic Research Consortium (BARC) 3-5 classified bleeding as in-patient, and up to 12 months
Stroke | 12 months
  Incidence of stroke
Cost effectiveness | 12 months
  Cost effectiveness of immediate PCI versus standard care
Left ventricular ejection fraction on cardiac MRI | 7 days (+/-3 days)
  Left ventricular ejection fraction on cardiac MRI
Infarct size on cardiac MRI | 7 days (+/-3 days)
  Infarct size on cardiac MRI
Proportion of patients needing emergency/urgent revascularisation | 3-4 days (standard of care timing angiography will vary between recruiting centres)
  Proportion of patients needing emergency/urgent revascularisation (in group B)
Total access site complications | 12 months
  Incidence of total VARC-2 classified access site complications as in-patient, and up to 12 months
Major access site complications | 12 months
  Incidence of major VARC-2 classified access site complications as in-patient, and up to 12 months
Sensitivity and specificity of novel biomarkers for predicting need for revascularisation | 3-4 days (standard of care timing angiography will vary between recruiting centres)
  Sensitivity and specificity of novel biomarkers in predicting which patients do or do not require PCI following diagnostic angiography

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Banning, Study Chair — Oxford University Hospitals NHS Trust
Locations (1):
- Glenfield Hospital, University Hospitals of Leicester NHS Trust, Leicester, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kite TA, Ladwiniec A, Greenwood JP, Gale CP, Anantharam B, More R, Hetherington SL, Khan SQ, O'Kane P, Rakhit R, Chase A, Barber S, Waheed G, Berry C, Flather M, McCann GP, Curzen N, Banning AP, Gershlick AH; RAPID NSTEMI Investigators. Very early invasive strategy in higher risk non-ST-elevation acute coronary syndrome: the RAPID NSTEMI trial. Heart. 2024 Mar 12;110(7):500-507. doi: 10.1136/heartjnl-2023-323513. PMID 38103913
- [Derived] Kite TA, Banning AS, Ladwiniec A, Gale CP, Greenwood JP, Dalby M, Hobson R, Barber S, Parker E, Berry C, Flather MD, Curzen N, Banning AP, McCann GP, Gershlick AH. Very early invasive angiography versus standard of care in higher-risk non-ST elevation myocardial infarction: study protocol for the prospective multicentre randomised controlled RAPID N-STEMI trial. BMJ Open. 2022 May 3;12(5):e055878. doi: 10.1136/bmjopen-2021-055878. PMID 35504645